CLINICAL TRIAL: NCT03966365
Title: Phase I Clinical Study, to Evaluate the Safety and Tolerability of the Preservative-free Ophthalmic Solution PRO-122 Compared With Krytantek Ofteno®, Elaborated by Sophia Laboratories, S.A. of C.V. on the Ocular Surface of Ophthalmologically and Clinically Healthy Subjects
Brief Title: Safety and Tolerability of the Preservative-free Ophthalmic Solution PRO-122 Compared With Krytantek Ofteno®
Acronym: PRO-122/I
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorios Sophia S.A de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SOPH122-0518/I
Record Dates: First submitted 2019-05-24; First posted 2019-05-29 (Actual); Results first posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Glaucoma
Keywords: Glaucoma; Krytantek; Krytantek PF; PRO-122
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Intervention Model Description: Phase I clinical trial, controlled, parallel group, double blind, randomized.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinding will correspond to the principal investigator and coinvestigator. In addition, the statistical analysis will be carried out in a blinded manner for the final analysis. Blinding can not be guaranteed in the subject.
  The masking will be done through the secondary container. The primary packaging will not be masked by the morphological difference between them. The sponsor and the research center will have two blind / non-blind teams.
  They will be identified by means of identical labels. Which, in accordance with current and applicable regulations, must contain at least:
  * Name, address and telephone number of the sponsor.
  * Pharmaceutical form and route of administration.
  * Lot Number.
  * Caption "Exclusively for clinical studies"
  * Date of Expiry
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRO-122 (Experimental): - Dosage: 1 drop every 12 hours, in both eyes
  Interventions: Drug: PRO-122
- Krytantek Ofteno® (Active Comparator): - Dosage: 1 drop every 12 hours, in both eyes
  Interventions: Drug: Krytantek Ofteno®

INTERVENTIONS:
Drug: PRO-122 — * PRO-122. Timolol 0.5% / brimonidine 0.2% / dorzolamide 2% ophthalmic solution free of preservatives. Prepared by Sophia Laboratories, S.A. of C.V., Zapopan, Jalisco, Mexico.
  * Route of administration: topical ophthalmic.
  Other Names: timolol 0.5%; brimonidine 0.2%; dorzolamide 2%; Krytantek PF; Krytantek Ofteno® Preservative Free
  Arms: PRO-122
Drug: Krytantek Ofteno® — * - 1. Krytantek Ofteno®. Timolol 0.5% / brimonidine 0.2% / dorzolamide 2% ophthalmic solution. Prepared by Sophia Laboratories, S.A. of C.V., Zapopan, Jalisco, Mexico.
  * - Route of administration: topical ophthalmic.
  Other Names: timolol 0.5%; brimonidine 0.2%; dorzolamide 2%
  Arms: Krytantek Ofteno®

SUMMARY:
Therapeutic indication: Ocular hypotensive Use: Primary open-angle glaucoma and ocular hypertension.

Objectives: To evaluate the safety and tolerability of the preservative-free formulation PRO-122 manufactured by Sophia Laboratories, S.A. of C.V. on the ocular surface of clinically healthy subjects.

Hypothesis: The ophthalmic solution PRO-122 presents a profile of safety and tolerability similar to Krytantek Ofteno®, in healthy subjects.

Methodology: Phase I clinical trial, controlled, parallel group, double blind, randomized.

Number of patients: n=24 12 subjects per group (both eyes). Main inclusion criteria:Clinically healthy subjects.

DETAILED DESCRIPTION:
Number of patients: n = 24 12 subjects per group (both eyes). Main inclusion criteria: Clinically healthy subjects.

Treatment duration: 7 days. Duration of subject in the study: 15 to 22 days.

Adverse events will be reported and cataloged based on the MedDRA dictionary and will be reported to the corresponding regulatory entity.

The sponsor will carry out monitoring or quality visits to the research sites where it corroborates the information of the source documents and will contrast them with the information presented in the electronic CRF. Electronic case report forms will be evaluated by the clinical research associate and the clinical team of the sponsor (medical ophthalmologist researcher and pharmacologist of clinical safety).

Statistical methodology:

The data will be expressed with measures of central tendency: mean and standard deviation for the quantitative variables. The qualitative variables will be presented in frequencies and percentages. The statistical analysis will be carried out by means of the Mann-Whitney U test for the quantitative variables for the difference between the groups. The difference between the qualitative variables will be analyzed by means of X2 (Chi2). An alpha ≤ 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* - Clinically healthy
* Ability to give your signed informed consent, and show willingness to comply with study procedures and to modify your lifestyle activities (Section 6.2.2)
* Age between 18 to 45 years.
* Indistinct sex.
* Women must ensure a hormonal contraceptive method or intrauterine device during the study period.
* Blood tests: within normal parameters or with a range of ± 20% as long as the subject is clinically healthy.

  * Blood count (BH): Hemoglobin, erythrocytes, hematocrit, total leukocytes, platelets, mean corpuscular volume and mean corpuscular hemoglobin.
  * Blood chemistry of three elements (QS): Glucose, urea and creatinine.
  * Liver function tests (PFH): Aspartate Aminotransferase and Alanine Aminotransferase, total bilirubin, direct and indirect.
* Visual ability 20/30 or better in both eyes.
* Vital signs within normal parameters.
* Intraocular pressure ≥10 and ≤ 21 mmHg.

Exclusion Criteria:

* Users of topical ophthalmic products of any kind.
* Users of medicines, or herbal products, by any other route of administration, with the exception of hormonal contraceptives in the case of women.
* Women who are pregnant or breastfeeding.
* Participation in clinical research studies 90 days prior to inclusion in the present study.
* Previous participation in this same study.
* Users of contact lenses.
* History of any chronic-degenerative disease.
* Inflammatory or infectious disease, active at the time of study entry.
* Injuries or traumatisms not resolved at the time of admission to the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leopoldo Baiza Durán, MD, Study Director — Laboratorios Sophia S.A de C.V.
Locations (1):
- Unidad Clínica de Bioequivalencia, S. de R.L. de C.V., Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Munoz-Villegas P, Navarro-Sanchez AA, Sanchez-Rios A, Olvera-Montano O, Baiza-Duran LM. Reexamining Ophthalmic Drugs, Safety and Tolerability in Phase 1 Clinical Trials. Ther Clin Risk Manag. 2021 Oct 21;17:1123-1134. doi: 10.2147/TCRM.S331294. eCollection 2021. PMID 34707360

RESULTS

PARTICIPANT FLOW:
Groups:
- PRO-122: - Dosage: 1 drop every 12 hours, in both eyes
  PRO-122: - PRO-122. Timolol 0.5% / brimonidine 0.2% / dorzolamide 2% ophthalmic solution free of preservatives. Prepared by Sophia Laboratories, S.A. of C.V., Zapopan, Jalisco, Mexico.
  - Route of administration: topical ophthalmic.
- Krytantek Ofteno®: - Dosage: 1 drop every 12 hours, in both eyes
  Krytantek Ofteno®: - - 1. Krytantek Ofteno®. Timolol 0.5% / brimonidine 0.2% / dorzolamide 2% ophthalmic solution. Prepared by Sophia Laboratories, S.A. of C.V., Zapopan, Jalisco, Mexico.
  - - Route of administration: topical ophthalmic.
Period: Overall Study
Arm/Group | PRO-122 | Krytantek Ofteno®
Started | 12 | 12
Completed | 11 | 12
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PRO-122 | Krytantek Ofteno® | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.1 (4.8) | 27.6 (6.8) | 26.3 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 7 | 6 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Latin | 12 | 12 | 24
Region of Enrollment [Count of Participants; unit: Participants]
  Mexico | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events
Description: primary security variable the adverse events will be evaluated with a scale of Present / Absent, it is a nominal variable, the normal value is absent. it will be evaluated by the number of reported cases per group.
Time Frame: during the 14 days of evaluation, including the safety call (day 14)
Population: The statistical analysis was by intention to treat (ITT)
Measure: Number; unit: adverse events
Arm/Group | PRO-122 | Krytantek Ofteno®
Number analyzed (Participants) | 12 | 12
adverse events | 28 | 31
Statistical Analysis 1: Comparison: PRO-122 vs Krytantek Ofteno®; Test type: Other; p = 0.706, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Eye Comfort Index
Description: It is a questionnaire designed to measure the irritation of the ocular surface with Rasch analysis to produce estimates on a linear scale of intervals (ratings: 0-100).The Eye comfort index contains items that focus on the discomfort associated with alterations of the ocular surface.
  Values closer or equal to one hundred (100) correspond to greater discomfort, while values closer or equal to zero (0) correspond to greater comfort.
Time Frame: will be evaluated at the end of the treatment, at the final visit (day 8)
Population: Analysis per protocol (PP)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PRO-122 | Krytantek Ofteno®
Number analyzed (Participants) | 12 | 12
units on a scale | 24.6 (12.6) | 27.0 (12.8)
Statistical Analysis 1: Comparison: PRO-122 vs Krytantek Ofteno®; Test type: Other; p = 0.622, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Number of Eyes With Epithelial Defects by Grade
Description: The epithelial defects will be evaluated by means of two stains, green lissamine and fluorescein, it is a discrete variable that will be realized by direct observation, it will be staged according to the degrees of the oxford scale that go from 0 to 5 (0-V) according to its severity, where 0 is the normal lower limit and 5 the upper limit of defects.
Time Frame: will be evaluated at the end of the treatment, at the final visit (day 8)
Population: The statistical analysis was per protocol (PP)
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | PRO-122 | Krytantek Ofteno®
Number analyzed (Participants) | 11 | 12
Number analyzed (eyes) | 22 | 24
eyes
  Green lissamine grade 0 | 20 | 16
  Green lissamine grade 1 | 2 | 4
  Green lissamine grade 2 | 0 | 4
  Green lissamine grade 3 | 0 | 0
  Green lissamine grade 4 | 0 | 0
  Fluorescein grade 0 | 22 | 22
  Fluorescein grade 1 | 0 | 2
  Fluorescein grade 2 | 0 | 0
  Fluorescein grade 3 | 0 | 0
  Fluorescein grade 4 | 0 | 0
Statistical Analysis 1: Comparison: PRO-122 vs Krytantek Ofteno®; Green lissamine treatment groups; Test type: Other; p = 0.081, Chi-squared, Corrected
Statistical Analysis 2: Comparison: PRO-122 vs Krytantek Ofteno®; Fluorescein treatment groups; Test type: Other; p = 0.490, Chi-squared, Corrected

4. Secondary Outcome: Visual Ability
Description: The visual capacity variable will be reported using as a unit of measure a fraction, this is taken from a visual test with the Snellen primer, it is a Nominal type variable. where the optimal vision is 20/20 or 1.0 in decimal and the worst 20/200 or 0.1 in decimal number.
  For the appropriate management of the data, the result of the fraction obtained from the snellen scale is transformed to decimals, in this case subjects close to or equal to 1.0 have better visual acuity while subjects close to or equal to 0.1 have worse visual acuity.
  The decimal equivalence scale is the result of the division of the fraction obtained in the Snellen chart. where 20/20 = 1.0; Do not confuse with Logmar scale where 20/20 = 0.0
  Equivalences Snellen Scale = decimals: 20/200=0.1, 20/100=0.2, 20/50=0.4, 20/40=0.5, 20/30=0.66, 20/25=0.8, 20/20=1.0, etc.
Time Frame: will be evaluated at the end of the treatment, at the final visit (day 8)
Population: the statistical analysis was per protocol (PP)
Measure: Mean (Standard Deviation); unit: Decimal score
Arm/Group | PRO-122 | Krytantek Ofteno®
Number analyzed (Participants) | 11 | 12
Decimal score | 0.949 (0.11) | 0.907 (0.14)
Statistical Analysis 1: Comparison: PRO-122 vs Krytantek Ofteno®; Test type: Other; p = 0.253, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Participants With Conjunctival Hyperemia (CH) by Grade
Description: Conjunctival hyperemia will be evaluated as an ordinal variable, by direct observation and staged using the Efron scale as Normal / Very Light / Mild / Moderate / Severe. Based on this scale, the normal and mild stages are considered without pathologies or normal. Mild, moderate and severe are considered pathological.
Time Frame: will be evaluated at the end of the treatment, at the final visit (day 8)
Population: the analysis was per protocol
Measure: Count of Participants; unit: Participants
Arm/Group | PRO-122 | Krytantek Ofteno®
Number analyzed (Participants) | 11 | 12
Participants
  Normal (0) | 10 | 9
  Very mild (1) | 0 | 3
  Mild (2) | 1 | 0
  Moderate (3) | 0 | 0
  Severe (4) | 0 | 0
Statistical Analysis 1: Comparison: PRO-122 vs Krytantek Ofteno®; Test type: Other; p = 0.031, Chi-squared, Corrected

6. Secondary Outcome: Participants With Chemosis
Description: The chemosis will be evaluated, as a nominal variable, by direct observation and it will be staged as present and absent, where the normality is that said variable is absent.
Time Frame: will be evaluated at the end of the treatment, at the final visit (day 8)
Population: the analysis was per protocol
Measure: Count of Participants; unit: Participants
Arm/Group | PRO-122 | Krytantek Ofteno®
Number analyzed (Participants) | 11 | 12
Participants | 0 | 0

7. Other Pre Specified Outcome: Changes in Intraocular Pressure
Description: the intraocular pressure will be evaluated by means of the Goldman applanation tonometry whose unit of measurement is millimeters of mercury (mmHg), it is a continuous variable and its normality range is between 11 - 21 mmHg
Time Frame: will be evaluated at the end of the treatment, at the final visit (day 8)
Population: the analysis was per protocol
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | PRO-122 | Krytantek Ofteno®
Number analyzed (Participants) | 11 | 12
mmHg | 12.32 (2.3) | 11.78 (1.8)
Statistical Analysis 1: Comparison: PRO-122 vs Krytantek Ofteno®; Test type: Other; p = 0.651, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored throughout the study, which lasted about 4 months.
Arm/Group | PRO-122 | Krytantek Ofteno®
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 11/12 | 11/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRO-122 (N=12) | Krytantek Ofteno® (N=12)
ocular burning (Eye disorders) | 11 (11) | 11 (11)
nonspecific conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
herpes labialis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
pruritus (Eye disorders) | 1 (1) | 2 (2)
ocular hyperemia (Eye disorders) | 2 (2) | 2 (2)
feeling of sticky eyes (Eye disorders) | 0 (0) | 1 (1)
decreased visual acuity (Eye disorders) | 1 (1) | 0 (0)
headache (Nervous system disorders) | 2 (2) | 1 (1)
rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
clogged ear (Ear and labyrinth disorders) | 1 (1) | 0 (0)
stomach ache (Gastrointestinal disorders) | 0 (0) | 1 (1)
foreign body sensation in eye (Eye disorders) | 0 (0) | 2 (2)
Dry Eye (Eye disorders) | 2 (2) | 1 (1)
eyestrain (Eye disorders) | 0 (0) | 3 (3)
dysgeusia (Gastrointestinal disorders) | 4 (4) | 0 (0)
tearing (Eye disorders) | 0 (0) | 2 (2)
dizziness (Gastrointestinal disorders) | 1 (1) | 0 (0)
earache (Ear and labyrinth disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
only the sponsor has the decision to disseminate or publish the information obtained from the investigation and the PIs involved must submit a formal request to the sponsor if they are willing to disseminate or publish such information, they may only publish them if they have the written authorization of the sponsor (Laboratoios Sophia S.A. de C.V.).

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-22): https://cdn.clinicaltrials.gov/large-docs/65/NCT03966365/Prot_SAP_000.pdf